CLINICAL TRIAL: NCT05410418
Title: A Phase II Study Evaluating the Efficacy of Mosunetuzumab in Combination With Polatuzumab Vedotin in Untreated Follicular Lymphoma
Brief Title: Mosunetuzumab and Polatuzumab Vedotin for Untreated Follicular Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Genentech, Inc. (Industry); Institute for Follicular Lymphoma (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202207147
Record Dates: First submitted 2022-05-26; First posted 2022-06-08 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Lymphoma, Follicular; Follicular Lymphoma
Keywords: lymphoma; follicular lymphoma; antibody-drug conjugate; B-NHL; B cell non-Hodgkin lymphoma; mosunetuzumab; polatuzumab vedotin; bispecific antibody
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma; Lymphoma, B-Cell | interventions — polatuzumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mosunetuzumab and Polatuzumab Vedotin (Experimental): Patients receive CD3xCD20 bispecific antibody mosunetuzumab administered subcutaneously in combination with CD79b directed ADC polatuzumab vedotin administered intravenously. Mosunetuzumab and polatuzumab vedotin are given in combination for 6 cycles. Mosunetuzumab is given on Days 1, 8, and 15 of cycle 1 and then Day 1 thereafter, and polatuzumab vedotin is given on Day 1. After 6 cycles, patients continue on mosunetuzumab alone for 2 additional cycles. Patients undergo scans at the end of cycle 8, and if those scans show a complete response, patients will stop any further treatment and will enter follow-up. Patients with a partial response or stable disease on scans at the end of cycle 8 may receive up to 9 additional cycles of mosunetuzumab in the absence of disease progression or unacceptable toxicity. All cycles are planned to be 21 days.
  Interventions: Drug: Mosunetuzumab; Drug: Polatuzumab vedotin

INTERVENTIONS:
Drug: Mosunetuzumab — Mosunetuzumab is administered subcutaneously using a "step-up" dosing strategy. The initial dose on C1D1 will be 5 mg, and doses thereafter will be 45 mg.
  Other Names: RO7030816; BTCT4465A
Drug: Polatuzumab vedotin — Polatuzumab vedotin is administered intravenously over 90 minutes for the initial dose, and over 30 minutes thereafter.
  Other Names: RO5541077; DCDS4501A

SUMMARY:
This phase II clinical trial studies the combination of mosunetuzumab and polatuzumab vedotin in order to see how well it works in patients with untreated follicular lymphoma. Mosunetuzumab is an antibody that has been engineered to attach to two target cells in the immune system: T cells that normally perform tasks like killing virus-infected cells, and cancerous B cells. Mosunetuzumab has been designed to direct these T cells to kill the cancerous B cells instead. Polatuzumab vedotin is an antibody-drug conjugate that attaches to certain cancerous B cells and then delivers a drug specifically to those cells.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of follicular lymphoma grade 1-3A, stage II-IV by Ann Arbor criteria.
* One or more of the following criteria (adapted from GELF criteria):

  * Any nodal or extranodal tumor mass with diameter > 7 cm
  * Involvement of at least 3 nodal sites, each with diameter > 3 cm
  * Presence of any systemic or B symptoms
  * Splenic enlargement with inferior margin below the umbilical line
  * Compression syndrome (e.g., ureteral, orbital, gastrointestinal)
  * Pleural or peritoneal serous effusion (irrespective of cell content)
  * Cytopenia(s) attributable to lymphoma
* At least 18 years of age.
* ECOG performance status ≤ 2
* Adequate hematologic and organ function (unless due to underlying lymphoma per the investigator; see below), defined as follows:

  * Absolute neutrophil count ≥ 1,000/mcL
  * Platelets ≥ 75,000/mcL
  * Hemoglobin ≥ 8 g/dL
  * Serum total bilirubin ≤ 1.5 x IULN (or ≤ 3 x IULN for patients with Gilbert syndrome)
  * AST(SGOT)/ALT(SGPT) ≤ 3 x IULN
  * Serum creatinine ≤ 1.0 x IULN or creatinine clearance ≥ 50 mL/min by Cockcroft-Gault
* Patients with extensive bone marrow involvement by lymphoma and/or disease-related cytopenias (e.g., immune thrombocytopenia) may be enrolled if the following criteria are met:

  * Absolute neutrophil count ≥ 500/mcL
  * Platelet count ≥ 50,000/mcL without platelet transfusion within 14 days prior to the first dose of mosunetuzumab
  * Hemoglobin ≥ 7 g/dL without red blood cell transfusion within 7 days prior to the first dose of mosunetuzumab
* The effects of mosunetuzumab on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study treatment, for 3 months following the final dose of mosunetuzumab, for 9 months after the final dose of polatuzumab vedotin, and for 3 months after the final dose of tocilizumab, as applicable. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study treatment, for 6 months after the final dose of polatuzumab vedotin, and for 2 months after the final dose of tocilizumab, as applicable.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Prior history of aggressive B cell lymphoma such as diffuse large B cell lymphoma or high-grade B cell lymphoma.
* Known history of treatment-emergent immune-related adverse events associated with prior immunotherapeutic agents.
* Known history of macrophage activation syndrome (MAS) or hemophagocytic lymphohistiocytosis (HLH).
* Current or past history of CNS lymphoma.
* Any prior systemic therapy for follicular lymphoma.
* Treatment with radiotherapy within 2 weeks prior to the first dose of mosunetuzumab (otherwise one measurable lesion outside of the radiation field must remain).
* Treatment with any anti-CD20 monoclonal antibody within 4 weeks of Day 1 of Cycle 1.
* Current or recent history (within the last 6 months) of CNS disease, such as stroke, epilepsy CNS vasculitis, or serious progressive neurodegenerative disease, with clinically significant symptoms.
* Treatment with systemic immunosuppressive medications, including but not limited to prednisone (> 20 mg), azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents within 2 weeks prior to Day 1 of Cycle 1.

  * Note: The use of inhaled corticosteroids, mineralocorticoids for management of orthostatic hypotension, and single dose dexamethasone for nausea or B symptoms is permitted.
* History of solid organ transplantation.
* History of allogeneic stem cell transplantation.
* Prior treatment with chimeric antigen receptor T cell therapy within 30 days before Day 1 of Cycle 1.
* History of severe allergic or anaphylactic reaction to humanized, chimeric, or murine monoclonal antibodies (mAbs).
* Known hypersensitivity to biopharmaceuticals produced in CHO cells or any component of the mosunetuzumab formulation, including mannitol.
* History of erythema multiforme, Grade ≥ 3 rash, or blistering following prior treatment with immunomodulatory derivatives.
* Known active bacterial, viral, fungal, or other infection, or any major episode of infection requiring treatment with IV antibiotics within 1 week of Day 1 of Cycle 1.
* Known or suspected chronic active Epstein-Barr virus (EBV) infection.
* Current Grade > 1 peripheral neuropathy by clinical examination or demyelinating form of Charcot-Marie-Tooth disease.
* Active hepatitis B infection.

  * Patients who are hepatitis B surface antigen (HBsAg) negative and hepatitis B core antibody (HBcAb) positive, must be negative for hepatitis B virus (HBV) polymerase chain reaction (PCR) to be eligible for study participation
* Active hepatitis C infection.

  * Patients who are positive for hepatitis C virus (HCV) antibody must be negative for HCV by PCR to be eligible for study participation
* Known history of human immunodeficiency virus (HIV) positive status.
* History of progressive multifocal leukoencephalopathy (PML).
* Administration of a live, attenuated vaccine within 4 weeks before first dose of study treatment or anticipation that such a live attenuated vaccine will be required during the study.

  * Patients must not receive live, attenuated vaccines (e.g., FluMist®) while receiving study treatment or after the last dose until B cell recovery to the normal ranges.
* Other malignancy that could affect compliance with the protocol or interpretation of results, with the exception of the following:

  * Any of the following malignancies previously curatively treated: carcinoma in situ of the cervix, good-prognosis ductal carcinoma in situ of the breast, basal, or squamous cell skin cancer
  * Stage I melanoma, low grade, early stage localized prostate cancer, or any other previously treated malignancy that has been in remission without treatment for at least 2 years prior to enrollment
* Active autoimmune disease requiring treatment.
* History of autoimmune disease, including, but not limited to, myocarditis, pneumonitis, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.

  * Patients with a remote history of, or well-controlled autoimmune disease, with a treatment free interval from immunosuppressive therapy for 12 months may be eligible to enroll if judged to be safe by the investigator.
  * Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid-replacement hormone are eligible.
  * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
  * Patients with a history of disease-related immune thrombocytopenic purpura, or autoimmune hemolytic anemia may be eligible.
* Evidence of any significant, uncontrolled concomitant disease that could affect compliance with the protocol or interpretation of results, including, but not limited to, significant cardiovascular disease (e.g., New York Heart Association Class III or IV cardiac disease, myocardial infarction within the previous 6 months, unstable arrhythmia, or unstable angina) or significant pulmonary disease (such as obstructive pulmonary disease or history of bronchospasm).
* Major surgical procedure other than for diagnosis within 28 days prior to Day 1 of Cycle 1 Day 1 or anticipation of a major surgical procedure during the course of the study.
* Pregnant or lactating or intending to become pregnant during the study.

  * Women of childbearing potential must have 1 negative serum pregnancy test result (minimum sensitivity, 25 mIU/mL) within 7 days of initiating Cycle 1 Day 1 of therapy.
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study, or which could affect compliance with the protocol or interpretation of results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2025-09-18 (Actual); Study Completion 2029-04-24 (Estimated)

PRIMARY OUTCOMES:
Number of participants with complete response (CR) as best response | Through completion of treatment (estimated to be 1 year)
  CR determined by response to treatment by PET-CT at end of treatment per Deauville 5-point scale (Lugano 2014 criteria). The Deauville scale is scored from 1 to 5, with 1 indicating no uptake on PET-CT and 5 indicating markedly increased uptake on PET-CT.

SECONDARY OUTCOMES:
Number of participants with complete response (CR) | After Cycle 8 (each cycle is 21 days; estimated to be 6 months)
  CR determined by response to treatment by PET-CT after Cycle 8 per Deauville 5-point scale (Lugano 2014 criteria). The Deauville scale is scored from 1 to 5, with 1 indicating no uptake on PET-CT and 5 indicating markedly increased uptake on PET-CT.
Number of participants with partial response (PR) | After Cycle 8 (each cycle is 21 days; estimated to be 6 months)
  PR determined by response to treatment by PET-CT after Cycle 8 per Deauville 5-point scale (Lugano 2014 criteria). The Deauville scale is scored from 1 to 5, with 1 indicating no uptake on PET-CT and 5 indicating markedly increased uptake on PET-CT.
Number of participants with partial response (PR) | Through completion of treatment (estimated to be 1 year)
  PR determined by response to treatment by PET-CT after Cycle 8 per Deauville 5-point scale (Lugano 2014 criteria). The Deauville scale is scored from 1 to 5, with 1 indicating no uptake on PET-CT and 5 indicating markedly increased uptake on PET-CT.
Overall response rate (ORR) as measured by number of participants with complete response (CR) and partial response (PR) | After Cycle 8 (each cycle is 21 days; estimated to be 6 months)
  CR and PR determined by response to treatment by PET-CT after Cycle 8 per Deauville 5-point scale (Lugano 2014 criteria). The Deauville scale is scored from 1 to 5, with 1 indicating no uptake on PET-CT and 5 indicating markedly increased uptake on PET-CT.
Overall response rate (ORR) as measured by number of participants with complete response (CR) and partial response (PR) | Through completion of treatment (estimated to be 1 year)
  CR and PR determined by response to treatment by PET-CT after Cycle 8 per Deauville 5-point scale (Lugano 2014 criteria). The Deauville scale is scored from 1 to 5, with 1 indicating no uptake on PET-CT and 5 indicating markedly increased uptake on PET-CT.
Number of participants with stable disease (SD) | After Cycle 8 (each cycle is 21 days; estimated to be 6 months)
  SD determined by response to treatment by PET-CT after Cycle 8 per Deauville 5-point scale (Lugano 2014 criteria). The Deauville scale is scored from 1 to 5, with 1 indicating no uptake on PET-CT and 5 indicating markedly increased uptake on PET-CT.
Number of participants with stable disease (SD) | Through completion of treatment (estimated to be 1 year)
  SD determined by response to treatment by PET-CT after Cycle 8 per Deauville 5-point scale (Lugano 2014 criteria). The Deauville scale is scored from 1 to 5, with 1 indicating no uptake on PET-CT and 5 indicating markedly increased uptake on PET-CT.
Number of participants with progressive disease (PD) | After Cycle 8 (each cycle is 21 days; estimated to be 6 months)
  PD determined by response to treatment by PET-CT after Cycle 8 per Deauville 5-point scale (Lugano 2014 criteria). The Deauville scale is scored from 1 to 5, with 1 indicating no uptake on PET-CT and 5 indicating markedly increased uptake on PET-CT.
Number of participants with progressive disease (PD) | Through completion of treatment (estimated to be 1 year)
  PD determined by response to treatment by PET-CT after Cycle 8 per Deauville 5-point scale (Lugano 2014 criteria). The Deauville scale is scored from 1 to 5, with 1 indicating no uptake on PET-CT and 5 indicating markedly increased uptake on PET-CT.
Number of participants with complete response (CR) | After Cycle 2 (each cycle is 21 days; estimated to be 42 days)
  CR determined by response to treatment by PET-CT after Cycle 2 per Deauville 5-point scale (Lugano 2014 criteria). The Deauville scale is scored from 1 to 5, with 1 indicating no uptake on PET-CT and 5 indicating markedly increased uptake on PET-CT.
Number of participants with partial response (PR) | After Cycle 2 (each cycle is 21 days; estimated to be 42 days)
  PR determined by response to treatment by PET-CT after Cycle 2 per Deauville 5-point scale (Lugano 2014 criteria). The Deauville scale is scored from 1 to 5, with 1 indicating no uptake on PET-CT and 5 indicating markedly increased uptake on PET-CT.
Overall response rate (ORR) as measured by number of participants with complete response (CR) and partial response (PR) | After Cycle 2 (each cycle is 21 days; estimated to be 42 days)
  CR and PR determined by response to treatment by PET-CT after Cycle 2 per Deauville 5-point scale (Lugano 2014 criteria). The Deauville scale is scored from 1 to 5, with 1 indicating no uptake on PET-CT and 5 indicating markedly increased uptake on PET-CT.
Number of participants with stable disease (SD) | After Cycle 2 (each cycle is 21 days; estimated to be 42 days)
  SD determined by response to treatment by PET-CT after Cycle 2 per Deauville 5-point scale (Lugano 2014 criteria). The Deauville scale is scored from 1 to 5, with 1 indicating no uptake on PET-CT and 5 indicating markedly increased uptake on PET-CT.
Number of participants with progressive disease (PD) | After Cycle 2 (each cycle is 21 days; estimated to be 42 days)
  PD determined by response to treatment by PET-CT after Cycle 2 per Deauville 5-point scale (Lugano 2014 criteria). The Deauville scale is scored from 1 to 5, with 1 indicating no uptake on PET-CT and 5 indicating markedly increased uptake on PET-CT.
Progression-free survival (PFS) | At 24 months
  Progression-free survival is defined from the time from study enrollment to the first occurrence of disease progression as determined by the investigator with use of the Lugano Response Criteria or death from any cause.
Progression-free survival (PFS) | At 48 months
  Progression-free survival is defined from the time from study enrollment to the first occurrence of disease progression as determined by the investigator with use of the Lugano Response Criteria or death from any cause.
Overall survival (OS) | At 24 months
  Overall survival is defined from the time from study enrollment to death from any cause.
Overall survival (OS) | At 48 months
  Overall survival is defined from the time from study enrollment to death from any cause.
Time to first response of complete response (CR) or partial response (PR) | Through completion of treatment (estimated to be 1 year)
  Response determined by PET-CT per the Deauville 5-point scale (Lugano 2014 criteria). The Deauville scale is scored from 1 to 5, with 1 indicating no uptake on PET-CT and 5 indicating markedly increased uptake on PET-CT. Response assessment is performed after cycle 2 (estimated to be day 42), after cycle 8 (estimated to be at 6 months), and at end of treatment (estimated to be 1 year).
Duration of first response of complete response (CR) or partial response (PR) | Through completion of treatment (estimated to be 1 year)
  Response determined by PET-CT per the Deauville 5-point scale (Lugano 2014 criteria). The Deauville scale is scored from 1 to 5, with 1 indicating no uptake on PET-CT and 5 indicating markedly increased uptake on PET-CT. Response assessment is performed after cycle 2 (estimated to be day 42), after cycle 8 (estimated to be at 6 months), and at end of treatment (estimated to be 1 year)
Time to first complete response (CR) | Through completion of treatment (estimated to be 1 year)
  Response determined by PET-CT per the Deauville 5-point scale (Lugano 2014 criteria). The Deauville scale is scored from 1 to 5, with 1 indicating no uptake on PET-CT and 5 indicating markedly increased uptake on PET-CT. Response assessment is performed after cycle 2 (estimated to be day 42), after cycle 8 (estimated to be at 6 months), and at end of treatment (estimated to be 1 year)
Duration of first complete response (CR) | Through completion of treatment (estimated to be 1 year)
  Response determined by PET-CT per the Deauville 5-point scale (Lugano 2014 criteria). The Deauville scale is scored from 1 to 5, with 1 indicating no uptake on PET-CT and 5 indicating markedly increased uptake on PET-CT. Response assessment is performed after cycle 2 (estimated to be day 42), after cycle 8 (estimated to be at 6 months), and at end of treatment (estimated to be 1 year)
Time to next treatment (TTNT) | Through completion of follow-up (estimated to be 6 years)
  Time to next treatment (TTNT) initiation is defined as the time from study enrollment to the first documented administration of a new anti-lymphoma treatment (including chemotherapy, radiotherapy, radioimmunotherapy, or immunotherapy) after completion of study treatment.
Frequencies and grades of treatment-emergent adverse events (TEAEs) | Evaluated from start of treatment to 30 day follow-up after conclusion of treatment, study discontinuation/termination, or initiation of alternative lymphoma-directed therapy, whichever occurs first (estimated to be 1 year and 30 days).
  TEAEs are defined as adverse events that are possibly, probably, or definitely related to study treatment and occur on or after first dose of study treatment..
Rate of treatment discontinuation due to treatment-emergent adverse events (TEAEs) | Evaluated from start of treatment to 30 day follow-up after conclusion of treatment, study discontinuation/termination, or initiation of alternative lymphoma-directed therapy, whichever occurs first (estimated to be 1 year and 30 days).
  TEAEs are defined as adverse events that are possibly, probably, or definitely related to study treatment and occur on or after first dose of study treatment..
Percentage of patients requiring any tocilizumab doses for management of cytokine release syndrome (CRS) | Up to approximately 1 year and 3 days
  Tocilizumab is recommended for treatment of grade 2 CRS and required for grade 3 or 4 CRS. Tocilizumab should be administered by IV infusion for a maximum of 4 doses.
Number of tocilizumab doses per patient for management of cytokine release syndrome (CRS) | Up to approximately 1 year and 3 days
  Tocilizumab is recommended for treatment of grade 2 CRS and required for grade 3 or 4 CRS. Tocilizumab should be administered by IV infusion for a maximum of 4 doses.

CONTACTS AND LOCATIONS:
Overall Officials: David A Russler-Germain, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu